CLINICAL TRIAL: NCT06010420
Title: The Effect of Using Medial Longitudinal Arch Supported Insoles on Jumping in Young Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Uskudar52
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Pes Planus; Sports Physical Therapy
Keywords: jumping; insoles; footballer
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: use of insoles
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- flat sole (Experimental): Weighted-unweighted in navicular drop test 10 mm or more pronation
  Interventions: Device: insoles
- normal base (Experimental): Weighted-unweighted in navicular drop test difference between measurement 5-9 mm is normal
  Interventions: Device: insoles
- high sole (Experimental): Weighted-unweighted in navicular drop test 4 mm or less is considered supination. are being
  Interventions: Device: insoles

INTERVENTIONS:
Device: insoles — Insoles are support devices that take the shape of the foot structure and enable the foot to press in a correct form.

SUMMARY:
In this study, it was aimed to determine the effect of pressing styles and insoles on jumping performances.

DETAILED DESCRIPTION:
In this clinical study, 30 healthy male football players between the ages of 16-20 will be carried out at Kasımpaşa Sports Club Academy. In the study, the effect of medial longitudinal arch height and the use of insoles on jumping using vertical jump, countermovement jump and drop jump tests will be investigated. Football players; Medial longitudinal arch heights will be measured by applying Foot Posture Index-6 and Navicular Position Test. As a result of these measurements; flat sole, normal sole and high sole will be divided into three groups. These three groups; Vertical jumping, countermovement jumping and drop jumping tests will be applied with the help of portable jumping apparatus and the results will be recorded. These tests will be re-applied to all three groups with a non-personalized, prefabricated insole that supports the medial arch. According to these tests, it will be investigated whether jumping performance depends on medial arch height. It will be evaluated whether there is a change in jumps after the insoles used. The obtained data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Football players between the ages of 16-20 will be included in the study.
* Football players who were not injured at the time of the study were included in the study will be.
* Football players who allow and want to participate in the study will be included in the study.

Exclusion Criteria:

• Football players who had an injury at the time of the study were included in the study will not be.

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Vertical jump test | 1 day
  It is a test used to determine the jump height in athletes. In our study; The jump starting position for this test will be with the knees flexed at 90 degrees, the head facing forward, the arms positioned freely at the side of the body. While jumping; Upward jumping will be required with a sudden thrust. During this jump, the ankle will be plantar flexed, the knees and hips extended, and the arms will be lifted upwards. During landing, the ankle will contact the ground with dorsiflexion, knees and hips extended, and return to the starting position. 3 repetitions will be done and the highest will be accepted.
Countermovement Jump Test | 1 day
  It is a frequently used method to evaluate the capacity of the musculoskeletal system in athletes. It is generally used to monitor the training capacity of athletes through parameters such as jump height, strength, power and speed. The jump start position for this test will be positioned with the knees flexed at 90 degrees, the head facing forward, with the hands on the waist from the sides to restrict the movement of the arms. While jumping; Upward jumping will be required with a sudden thrust. During this jump, the ankle will be plantar flexed, the knees and hips will be extended, and the hands will be at the waist. During landing, the ankle will contact the ground with dorsiflexion, knees and hips extended, and return to the starting position. 3 repetitions will be done and the highest will be accepted.
Drop Jump Test | 1 day
  In our study, the starting position for this test will be on a high jump box with the hands at the sides on the waist and in a standing upright position. To initiate the fall movement, participants will be instructed: "step out of the box with one foot and try to make the highest jump immediately after contact with the ground". The player will be instructed not to leave the jumping platform and jump out of the box for landing and jumping. The jump box will be 30 cm high. 3 repetitions will be done and the highest will be accepted. Reliability tests were conducted for jumping tests.
Navicular position test | 1 day
  The test is done standing up. For whichever foot it will be applied, that foot will be in the back, the other foot will be in front, and the calcaneus of the front foot and the tip of the toe of the back foot will be on the same horizontal plane. In the extremity to be applied, the knee will be kept in a bent position so that it is vertically aligned with the 1st and 2nd finger. In this position, mark the head of the 1st metatarsal bone, the navicular bone, the apex of the medial malleolus, and the dorsal of the Achilles tendon horizontally aligned. First, a line is drawn and extended between the head of the 1st metatarsal bone and the navicular bone. Second, a line is drawn and lengthened between the navicular bone and the Achilles tendon. The angle between these two lines is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Can GÜNGÖRDÜ, Study Chair — Kasimpasa Sports Club
Locations (1):
- Kasimpasa Sports Club, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brocherie F, Millet GP, Girard O. Neuro-mechanical and metabolic adjustments to the repeated anaerobic sprint test in professional football players. Eur J Appl Physiol. 2015 May;115(5):891-903. doi: 10.1007/s00421-014-3070-z. Epub 2014 Dec 7. PMID 25481506
- [Background] Madeleine P, Hoej BP, Fernandez-de-Las-Penas C, Rathleff MS, Kaalund S. Pressure pain sensitivity changes after use of shock-absorbing insoles among young soccer players training on artificial turf: a randomized controlled trial. J Orthop Sports Phys Ther. 2014 Aug;44(8):587-94. doi: 10.2519/jospt.2014.5117. Epub 2014 Jul 16. PMID 25029914
- [Background] Girard O, Millet GP, Thomson A, Brocherie F. Is Plantar Loading Altered During Repeated Sprints on Artificial Turf in International Football Players? J Sports Sci Med. 2018 Aug 14;17(3):359-365. eCollection 2018 Sep. PMID 30116108
- [Background] Arundale AJH, Kvist J, Hagglund M, Faltstrom A. Jump performance in male and female football players. Knee Surg Sports Traumatol Arthrosc. 2020 Feb;28(2):606-613. doi: 10.1007/s00167-019-05747-1. Epub 2019 Oct 30. PMID 31667569
- [Background] Loturco I, Jeffreys I, Abad CCC, Kobal R, Zanetti V, Pereira LA, Nimphius S. Change-of-direction, speed and jump performance in soccer players: a comparison across different age-categories. J Sports Sci. 2020 Jun-Jun;38(11-12):1279-1285. doi: 10.1080/02640414.2019.1574276. Epub 2019 Feb 6. PMID 30724662